CLINICAL TRIAL: NCT06645756
Title: Comparative Analysis of Postprandial Effects in Healthy and Obese Individuals
Acronym: CAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UniHohMet-CAPE-2023
Record Dates: First submitted 2023-09-21; First posted 2024-10-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Normal Weigth
Keywords: high-fat diet; high-calorie diet; leukocytes; LPS
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obese group (Experimental): Test meal
  Interventions: Other: Test meal
- Normal weight group (Experimental): Test meal
  Interventions: Other: Test meal

INTERVENTIONS:
Other: Test meal — Test meal consisting of fries, chicken nuggets and eggs

SUMMARY:
After eating, blood composition changes, including increased triglycerides and glucose, which can trigger postprandial inflammation. Particularly with high-fat foods, pro-inflammatory lipopolysaccharide (LPS) increases. This activates leukocytes to release pro-inflammatory cytokines. In industrialized countries where "snacking" is common, many people spend the day in a postprandial state. Obese individuals tend to have chronic inflammation and show increased susceptibility to infections such as SARS-CoV-2. The main objective of the study is to investigate the response of leukocytes and the serum metabolome after food intake in individuals with obesity compared to healthy individuals, focusing on LPS as a key stimulus of innate immunity.

ELIGIBILITY:
Inclusion Criteria:

* Signed declaration of consent
* from 25 years of age
* BMI 20 kg/m2 - 25 kg/m2 or BMI 30 kg/m2 - 40 kg/m2
* Good venous conditions for blood collection
* Sufficient understanding of the German language and sufficient mental state to understand information and instructions related to the study

Exclusion Criteria:

* Nicotine consumption
* High-risk alcohol consumption (more than one standard glass per day for women, more than two standard glasses per day for men)
* Antibiotic intake
* Taking probiotics, prebiotics and synbiotics, unless taken for more than 90 days
* Taking statins or other lipid-lowering medications (e.g., ezetimibe, fibrates)
* Taking oral antidiabetics
* Taking antacids
* Manifest diabetes mellitus
* Acute/unstable cardiovascular diseases
* Acute inflammatory diseases
* autoimmune diseases
* kidney diseases
* food allergy or food intolerance to food components of the test meal (e.g. eggs)
* celiac disease
* Pregnancy and lactation
* Inability to consume the test meal orally
* Placement in a clinic or similar facility due to official or court order (medical history)
* Participation in another clinical study (current or within the last 30 days prior to study entry)
* A medical condition or regular medication use that, at the investigator's discretion, does not permit study participation or evaluation of study parameters or consumption of the investigational product (individual decision)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
LPS | 30 min after test meal
  LPS in Serum
LPS | 60 min after test meal
  LPS in Serum
LPS | 120 min after test meal
  LPS in Serum
LPS | 180 min after test meal
  LPS in Serum
LPS | 240 min after test meal
  LPS in Serum

SECONDARY OUTCOMES:
Activability of PBMCs in vitro | immediately after the intervention
  To analyze the reactivity of PBMCs, these are isolated, co-cultivated with bacteria and then the number of replicable bacteria is counted.
Serum cytokines and PAMPs | immediately after the intervention
Characterization of PBMCs | immediately after the intervention
  The PBMCs are characterized by fluorescence-activated cell sorting (FACS) and RNA isolation.
Metabolome analyses | immediately after the intervention
Trimethylamine / SCFA in serum | immediately after the intervention
Fasting blood glucose | immediately after the intervention
lipoproteins | immediately after the intervention
HbA1c | immediately after the intervention

OTHER OUTCOMES:
Microbiome RNA in serum | baseline
IgA in serum | immediately after the intervention
Fecal microbiome analysis | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Professor, Principal Investigator — University of Hohenheim
Locations (1):
- Metabolic Unit der Universität Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Case-by-case decision after contact